CLINICAL TRIAL: NCT02747602
Title: A Phase 1, Pilot, Single-Dose, 3-Way Crossover Study to Evaluate the Pharmacokinetic of AC-1204 Versus Caprylic Triglyceride Oil Including the Effect of Food on Ketone Body Production
Brief Title: Evaluation of PK of AC1204 v Caprylic Triglyceride Oil Incl Food Effect on Ketone Body Production
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cerecin (Industry)
Collaborators: Celerion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: AC-16-011_BE
Record Dates: First submitted 2016-04-15; First posted 2016-04-22 (Estimated); Last update posted 2016-10-28 (Estimated); Status verified 2016-10

CONDITIONS: Healthy
Keywords: Healthy volunteers; Caprylic triglyceride oil; AC-1204; Pharmacokinetic; Ketone body
MeSH Terms: interventions — tricaprylin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group ABC (Experimental): AC-1204, caprylic triglyceride oil standard breakfast, caprylic triglyceride high fat breakfast
  Interventions: Drug: AC-1204; Drug: caprylic triglyceride oil (standard breakfast); Drug: caprylic triglyceride oil (high fat breakfast)
- Group BCA (Experimental): caprylic triglyceride oil standard breakfast, caprylic triglyceride high fat breakfast, AC-1204
  Interventions: Drug: AC-1204; Drug: caprylic triglyceride oil (standard breakfast); Drug: caprylic triglyceride oil (high fat breakfast)
- Group CAB (Experimental): caprylic triglyceride high fat breakfast, AC-1204, caprylic triglyceride oil standard breakfast
  Interventions: Drug: AC-1204; Drug: caprylic triglyceride oil (standard breakfast); Drug: caprylic triglyceride oil (high fat breakfast)

INTERVENTIONS:
Drug: AC-1204 — 40 g (120 mL) AC-1204 administered 30 minutes after the start of a standard breakfast.
Drug: caprylic triglyceride oil (standard breakfast) — 20 g CT oil (21 mL) administered 30 minutes after the start of a standard breakfast.
Drug: caprylic triglyceride oil (high fat breakfast) — 20 g CT oil (21 mL) administered 30 minutes after the start of a high fat breakfast.

SUMMARY:
To compare serum ketone body (i.e., total ketones and β-hydroxybutyrate) levels after administration of AC-1204 versus caprylic triglyceride (CT) oil, both after a standard breakfast.

To evaluate the effect of a high fat diet on serum ketone body levels after administration of CT oil with a high fat breakfast versus a standard breakfast.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy, adult, male 18-55 years of age, inclusive, at screening.
2. Continuous non-smoker who has not used nicotine-containing products for at least 3 months prior to the first dose and throughout the study.
3. Body mass index (BMI) ≥ 20.0 and ≤ 30.0 kg/m2 at screening.
4. Medically healthy with no clinically significant medical history, physical examination, laboratory profiles, vital signs or ECGs, as deemed by the PI or designee. At screening, subjects must have alanine aminotransferase (ALT), aspartate aminotransferase (AST) and alkaline phosphatase (ALP) < the upper limit of normal and triglycerides levels < 250 mg/dL.
5. A non-vasectomized subject must agree to use a condom with spermicide or abstain from sexual intercourse during the study until 90 days beyond the last dose of study drug. (No restrictions are required for a vasectomized male provided his vasectomy has been performed 4 months or more prior to first dose/dosing of study drug. A subject who has been vasectomized less than 4 months prior to study first dose/dosing must follow the same restrictions as a non-vasectomized male).
6. Subjects must agree not to donate sperm from the first dose/dosing until 90 days after dosing.
7. Understands the study procedures in the informed consent form (ICF), and be willing and able to comply with the protocol.

Exclusion Criteria:

1. Subject is mentally or legally incapacitated or has significant emotional problems at the time of the screening visit or expected during the conduct of the study.
2. History or presence of clinically significant medical or psychiatric condition or disease in the opinion of the PI or designee.
3. History of any illness that, in the opinion of the PI or designee, might confound the results of the study or poses an additional risk to the subject by their participation in the study.
4. History or presence of alcoholism or drug abuse within the past 2 years prior to the first dose/dosing.
5. History or presence of hypersensitivity or idiosyncratic reaction to the study drugs, related compounds, milk, coconut oil, or soy.
6. History or presence of diverticular disease, ulcers, inflammatory bowel disease or recurrent diarrhea or gout.
7. Positive urine drug or alcohol results at screening or check-in.
8. Positive results at screening for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg) or hepatitis C virus (HCV).
9. Seated blood pressure is less than 90/40 mmHg or greater than 140/90 mmHg at screening.
10. Seated heart rate is lower than 40 bpm or higher than 99 bpm at screening.
11. QTc interval is >460 msec (males) or has ECG findings deemed abnormal with clinical significance by the PI or designee at screening.
12. Estimated creatinine clearance ≤80 mL/min at screening.
13. Unable to refrain from or anticipates the use of any drug, including prescription and non-prescription medications, herbal remedies, or vitamin supplements beginning 14 days prior to the first dose and throughout the study. Acetaminophen (up to 2 g per 24 hour period) and medications for the treatment of adverse events may be permitted during the study.
14. Has been on a diet incompatible with the on-study diet, in the opinion of the PI or designee, within the 28 days prior to the first dose and throughout the study.
15. Is lactose intolerant.
16. Is unable to complete the critical meal (i.e., breakfast prior to dosing).
17. Donation of blood or significant blood loss within 56 days prior to the first dose.
18. Plasma donation within 7 days prior to the first dose.
19. Participation in another clinical study within 28 days prior to the first dose. The 28-day window will be derived from the date of the last blood collection or dosing, whichever is later, in the previous study to Day 1 of Period 1 of the current study.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2016-04; Primary Completion 2016-05 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
total ketones AUC0-t | 0-24 hours
  The area under the concentration-time curve, from time 0 to the last observed non-zero concentration, as calculated by the linear trapezoidal method.
total ketones AUC0-inf | 0-24 hours
  The area under the concentration-time curve from time 0 extrapolated to infinity. AUC0-inf is calculated as the sum of AUC0-t plus the ratio of the last measurable serum concentration to the elimination rate constant.
total ketones AUC%extap | 0-24 hours
  Percent of AUCo-inf extrapolated, represented as (1 - AUC0-t/AUC0- inf)*100
total ketones Cmax | 0-24 hours
  Maximum observed concentration
total ketones Kel | 0-24 hours
  Apparent first-order terminal elimination rate constant calculated from a semi-log plot of the serum concentration versus time curve. The parameter will be calculated by linear least-squares regression analysis using the maximum number of points in the terminal log-linear phase (e.g., three or more non-zero serum concentrations)
total ketones T 1/2 | 0-24 hours
  Apparent first-order terminal elimination half-life will be calculated as 0.693/Kel
total ketones Tmax | 0-24 hours
  Time to reach Cmax. If the maximum value occurs at more than one time point, Tmax is defined as the first time point with this value
β-hydroxybutyrate AUC0-t | 0-24 hours
  The area under the concentration-time curve, from time 0 to the last observed non-zero concentration, as calculated by the linear trapezoidal method.
β-hydroxybutyrate AUC0-inf | 0-24 hours
  The area under the concentration-time curve from time 0 extrapolated to infinity. AUC0-inf is calculated as the sum of AUC0-t plus the ratio of the last measurable serum concentration to the elimination rate constant
β-hydroxybutyrate AUC%extap | 0-24 hours
  Percent of AUCo-inf extrapolated, represented as (1 - AUC0-t/AUC0- inf)*100.
β-hydroxybutyrate Cmax | 0-24 hours
  Maximum observed concentration
β-hydroxybutyrate Tmax | 0-24 hours
  Time to reach Cmax. If the maximum value occurs at more than one time point, Tmax is defined as the first time point with this value
β-hydroxybutyrate Kel | 0-24 hours
  Apparent first-order terminal elimination rate constant calculated from a semi-log plot of the serum concentration versus time curve. The parameter will be calculated by linear least-squares regression analysis using the maximum number of points in the terminal log-linear phase (e.g., three or more non-zero serum concentrations).
β-hydroxybutyrate T 1/2 | 0-24 hours
  Apparent first-order terminal elimination half-life will be calculated as 0.693/kel.

CONTACTS AND LOCATIONS:
Overall Officials: Geri Poss, MD, Principal Investigator — Celerion
Locations (1):
- Celerion, Inc, Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: No